CLINICAL TRIAL: NCT03207217
Title: Virtual Training Role-Plays to Improve Patient Suicide Outcomes in Primary Care Settings
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SIMmersion, LLC (Industry)
Collaborators: The Institute for Family Health (Other); Education Development Center, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R44MH114710-01 (NIH)
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Suicidal Ideation
Keywords: Safety Planning; Access to Lethal Means; Zero Suicide
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase I Knowledge Assessment (Experimental)
  Interventions: Other: Web-based training Product
- Phase II Efficacy (Experimental)
  Interventions: Other: Web-based training Product
- Phase II Acceptability (Experimental)
  Interventions: Other: Web-based training Product

INTERVENTIONS:
Other: Web-based training Product — A series of 4 modules to train providers to more effectively manage patients who screen positive for risk of suicide. The modules are: Risk Assessment, Safety Planning, Access to Lethal Means, and Willingness to accept referral.

SUMMARY:
SIMmersion, in collaboration with the Institute for Family Health (IFH) and the Educational Development Center (EDC) propose to develop a web-based training product, Suicide Prevention Role-plays for Interactive Training (SPiRIT), a series of 4 modules to train providers to more effectively manage patients who screen positive for risk of suicide in this Phase I/Phase II fast-track application. If funded, the team will develop the Risk Assessment module in Phase I and utilize a within group pre-post design to evaluate its feasibility. Twenty practicing clinicians will be recruited to utilize the module and complete a pre-post knowledge test. In Phase II, the team will develop Safety Planning, Access to Lethal Means, and Willingness to Accept a Referral modules. The efficacy of the product to positively influence patient outcomes will be tested with a Historically Controlled Trial (HCT) enlisting 65 practicing clinicians across five IFH sites. All providers will be trained and patient outcomes will be tracked for 6 months post training. This data set will be compared to 6 months of historical data for the same provider group. Primary outcomes of this study will measure the participants' ability in obtain improved patient outcomes related to: 1) rate of same-day C-SSRS Screening; 2) rate of suicide being added to the problem list; 3) rate of same-day safety planning; 4) rate of same day C-SSRS Lifeline/Recent Completion; 5) rate of same-day Risk Assessment; 6) rate of acceptance and attendance to within-Institute referrals for post intervention patients who are offered the referral at the first visit; 7) and lower rates of documented suicide attempts. Ultimately, the development and successful testing of this product would provide the US health care system a novel technology to scale up a clinician's confidence and skill to better manage patients who identify as at-risk for suicide. Additionally, if effective, this product will have a direct impact on patient outcomes, a vital component to any training product that attempts to train health care professionals. The utility and scalability of the proposed product will move health care systems toward the goal of zero deaths from suicide consistent with the Zero suicide approach.

ELIGIBILITY:
Inclusion Criteria:

(1) Hold an active license issued by the State of New York for their profession and be in good standing; (2) actively see patients at an IFH site; and (3) have completed IFH's mandated suicide prevention training.

Exclusion Criteria:

(1) have not completed their IFH Suicide Prevention Training as outlined in the IFH's Suicide Prevention Training Policy; or (2) have uncorrected vision or hearing problems that prevent the person from using the software. Specific to Phase II an additional criteria is (3)participated in the Phase 1 feasibility testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
C-SSRS Screening | Assessment will occur after a 6 month period of tracking patient records for each provider
  Higher rates of same-day C-SSRS Screening
Suicide addition to Problem List | Assessment will occur after a 6 month period of tracking patient records for each provider
  Higher rates of suicide being added to the problem list
Same-day Safety Planning, if a positive screen | Assessment will occur after a 6 month period of tracking patient records for each provider
  Higher rates of same-day Safety Planning, if a positive screen
C-SSRS Lifeline/Recent Completion | Assessment will occur after a 6 month period of tracking patient records for each provider
  Higher rates of same-day C-SSRS Lifeline/Recent Completion, if a positive screen;
Risk Assessment | Assessment will occur after a 6 month period of tracking patient records for each provider
  Higher rates of same-day Risk Assessment, if a positive screen
Within-Institute referrals | Assessment will occur after a 6 month period of tracking patient records for each provider
  Higher rates of acceptance and attendance to within-Institute referrals for post intervention patients who are offered the referral at the first visit
Documented suicide attempts | Assessment will occur after a 6 month period of tracking patient records for each provider
  Have lower rates of documented suicide attempts